CLINICAL TRIAL: NCT02992301
Title: Assessment of Atherosclerotic Plaque Characteristics Change by DCE-MRI With Alirocumab - a Pilot Study
Brief Title: Assessment of Atherosclerotic Plaque Characteristics Change by DCE-MRI With Alirocumab
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Westside Medical Associates of Los Angeles (Other)
Collaborators: University of Washington (Other); Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Norman Lepor, MD, Principal Investigator, Westside Medical Associates of Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WMALA-99-032
Record Dates: First submitted 2016-11-30; First posted 2016-12-14 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Atherosclerosis; Hyperlipidemia
MeSH Terms: conditions — Atherosclerosis; Hyperlipidemias | interventions — alirocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label (Experimental): All enrolled patients will receive open label Praluent (Alirocumab).
  Interventions: Drug: Alirocumab

INTERVENTIONS:
Drug: Alirocumab — Injectable prescription medicine called a PCSK9 inhibitor.
  Other Names: Praluent

SUMMARY:
Aim 1: To determine whether therapy with Alirocumab, compared to pre-treatment, will effectively improve carotid atherosclerotic plaque characteristics by reducing Ktrans and LRNC size. To achieve this goal, we will (a) enroll 30 subjects who are intolerant to high intensity statin therapy and only able to tolerate low potency statin or low weekly dose of high potency statin and have LDL-C ≥70 mg/dl; (b) initiate alirocumab at 150mg subcutaneously injection every 2 weeks; (c) perform carotid DCE-MRI scans at baseline, 3, 6 and 12 months; (d) perform quantitative analysis for vascular inflammation and plaque LRNC volume and other plaque characteristics; (e) compare vascular inflammation and LRNC volume between pre- and post-alirocumab at 3, 6 and 12 months.

Aim 2: To examine associations between reductions in atherogenic lipids (LDL-C, Lp(a), non-HDL-C) and changes in atherosclerotic plaque characteristics. To achieve this goal, we will (a) perform laboratory assessments of lipids, lipoproteins and apo-lipoproteins at baseline and during the study; (b) compare lipids, lipoproteins and apo-lipoproteins levels between pre- and post-alirocumab; (c) correlate reductions in atherogenic lipids with changes atherosclerotic plaque characteristics.

DETAILED DESCRIPTION:
Acute ischemic events caused by atherosclerosis cardiovascular disease (ASCVD) are primarily due to plaque rupture/erosion determined by plaque morphologic characteristics, local composition and inflammation, which can be directly assessed using magnetic resonance imaging (MRI). Prospective carotid MRI studies have demonstrated: (1) plaques with thin or ruptured cap, intraplaque hemorrhage (IPH), neovascularization, or larger lipid-rich necrotic core (LRNC) are strongly associated with occurrence of cerebrovascular and coronary events, (2) increased LRNC size is significantly associated with increased risk for systemic ASCVD events after adjusting for LDL-C or Non-HDL-C levels, (3) increased permeability of adventitial vasa vasorum is associated with presence of IPH which increases plaque burden and LRNC progression that appears to be resistant to conventional doses of statins, (4) intensive lipid therapy decreases carotid LRNC and vascular inflammation, (5) multicenter carotid studies can be conducted with good reproducibility and feasibility.

Unlike previous clinical trials evaluating carotid artery disease using ultrasound based technology that showed a weak relationship to systemic and coronary vascular events, recent studies have demonstrated predictive value of carotid plaque tissue characteristics for subsequent systemic ASCVD events including coronary events. Hellings and colleagues found that carotid plaque composition by histology in 818 patients who underwent endarterectomy is an independent predictor of future cardiovascular events during long-term post-operative follow-up. Specifically, those with carotid IPH and increased neovascularization were at significantly higher risk for ASCVD events. The Atherosclerosis Risk in Communities study investigators reported that carotid LRNC (HR=1.9, p=0.014) and minimum cap thickness (HR=0.67, p=0.03), as identified by MRI, were significantly associated with development of ASCVD including coronary events after adjusting for all clinical risk factors, treatment variables and biomarkers. The carotid MRI sub-study in AIM-HIGH showed that higher Lp(a) levels are associated with high-risk plaque features which are prevalent in subjects with established vascular disease and "well-controlled" LDL-C and blood pressure. Thin or ruptured cap and a larger LRNC are predictive of systemic ASCVD events that include 83% (15/18) of the coronary events in AIM-HIGH, meanwhile, none of the clinical risk factors and lipids were predictive of future events.

Alirocumab has shown substantial lowering in LDL-C, non-HDL-C and Lp(a), with or without concomitant statin treatment [43]. It has the potential to be a therapy that can improve plaque characteristics leading to reduction of ASCVD events. We propose to conduct a carotid MRI pilot study to demonstrate that adding alirocumab for 12 months, in comparison to pre-alirocumab therapy, in 30 subjects with documented carotid artery plaques who are not able to tolerate high intensity statin therapy and have LDL-C ≥70 mg/dl would improve atherosclerotic plaque characteristics by reducing Ktrans and LRNC size.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years of age.
* Subjects with documented inability to consistently take or tolerate high intensity statin therapy and LDL-C ≥70 mg/dL.
* Subjects are only able or allowed to take lower potency statin or low weekly dose of high potency statin due to concern of drug-to-drug interactions or lack of tolerance (pravastatin ≤140 mg, pitavastatin ≤14 mg, simvastatin ≤140 mg, atorvastatin ≤70 mg, or rosuvastatin ≤70 mg, weekly) or intolerant of all statin doses and with fasting LDL-C ≥100 mg/dL.
* Subjects must have significant carotid artery plaque with maximum wall thickness ≥2 mm on ultrasound performed within twelve months of screening.
* Subject must present with a LRNC on baseline MRI scan.
* Subjects must show an adequate image quality for MRI analysis.
* Medically stable.
* Willing to participate and sign informed consent.

Exclusion Criteria:

* Contraindication to MRI.
* Have immediate plans for bilateral carotid endarterectomy.
* Had received 2 or more doses of treatment with a PCSK9 inhibitor in the past 4 months.
* GFR ≤45 mL/min/1.73 m2 prior to MRI scan.
* Claustrophobia.
* Pregnant women; breastfeeding women; men and women of childbearing potential who are unwilling or unable to use a highly effective method of contraception.
* TIA or stroke within the preceding twelve months
* Severe carotid stenosis in an asymptomatic patient defined as any one of the following:

  1. Greater than or equal to 70% luminal narrowing on any imaging modality
  2. Peak systolic velocity greater than or equal to 250 cm/second
  3. End diastolic velocity greater than or equal to 100 cm/second
  4. Systolic volume ratio greater than or equal to 3.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Changes in carotid atherosclerotic plaque characteristics as evidenced by effect on the volume transfer constant( Ktrans) and lipid-rich necrotic core (LRNC) size. | 52 weeks
  To determine whether therapy with Alirocumab, compared to pre-treatment, will effectively improve carotid atherosclerotic plaque characteristics by reducing Ktrans and LRNC size. To achieve this goal, we will (a) enroll 30 subjects who are intolerant to high intensity statin therpay and only able to tolerate low potency statin or low weekly dose of high potency statin and have LDL-C ≥100 mg/dl; (b) initiate alirocumab at 150mg subcutaneously injection every 2 weeks; (c) perform carotid DCE-MRI scans at baseline, 3, 6 and 12 months; (d) perform quantitative analysis for vascular inflammation (Ktrans) and plaque LRNC volume and other plaque characteristics; (e) compare Ktrans and LRNC volume between pre- and post-alirocumab at 3, 6 and 12 months.

SECONDARY OUTCOMES:
Associations between reductions in atherogenic lipids and changes in atherosclerotic plaque characteristics | 52 weeks
  To examine associations between reductions in atherogenic lipids (LDL-C, Lp(a), non-HDL-C) and changes in atherosclerotic plaque characteristics. To achieve this goal, we will (a) perform laboratory assessments of lipids, lipoproteins and apo-lipoproteins at baseline and during the study; (b) compare lipids, lipoproteins and apo-lipoproteins levels between pre- and post-alirocumab; (c) correlate reductions in atherogenic lipids with changes atherosclerotic plaque characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Lepor, MD, Principal Investigator — Westside Medical Associates of Los Angeles
Locations (1):
- Westside Medical Associates of Los Angeles, Beverly Hills, California, United States

IPD SHARING:
Plan to Share IPD: Undecided